CLINICAL TRIAL: NCT07257172
Title: Sutureless Technique for Repositioning and Scleral Fixation of the Capsular Bag - Intraocular Lens Complex With Permanent Use of Iris Retractors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12/WIM/2021
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Lens Subluxation
Keywords: Lens Subluxation; iris retractors; sutureless fixation
MeSH Terms: conditions — Lens Subluxation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scleral fixation of the capsular bag-intraocular lens complex with permanent use of iris retractors (Experimental): Scleral fixation of the capsular bag-intraocular lens complex with permanent use of iris retractors
  Interventions: Procedure: Sutureless technique for repositioning and scleral fixation of the capsular bag - intraocular lens complex with permanent use of iris retractors

INTERVENTIONS:
Procedure: Sutureless technique for repositioning and scleral fixation of the capsular bag - intraocular lens complex with permanent use of iris retractors — The surgery was performed under retrobulbar anesthesia with 2% xylocaine and 0.5% bupivacaine. A 2.2 mm temporal clear-corneal incision and three side ports were created, followed by capsulorhexis with forceps. Due to limited vitreous prolapse, anterior vitrectomy was required. Iris retractors were inserted through the ports and positioned under the anterior capsule at the site of zonular loss. Phacoemulsification was completed with standard or reduced flow, a CTR was implanted, and a foldable one-piece IOL was placed in the bag. After removing the silicone stoppers, the retractors were lifted from the capsulotomy. A 25-gauge needle was passed 2 mm posterior to the limbus into the anterior chamber, aligned with zonular damage. The tip of one retractor was inserted into the needle and externalized; the ends were trimmed, cauterized, and the melted tip fixed subconjunctivally.

SUMMARY:
Sutureless technique for repositioning and scleral fixation of the capsular bag-intraocular lens complex with permanent use of iris retractors

DETAILED DESCRIPTION:
Purpose of the study is to present results of sutureless technique for repositioning and scleral fixation of the capsular bag-intraocular lens (IOL) complex in the surgical treatment of subluxated lenses. The investigators rated the BCVA, refractive outcomes, intraocular pressure, , tilt and decentration, and also determined intra- and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* only adult men and women with subluxation lens

Exclusion Criteria:

* previous ocular surgery
* Fuchs' dystrophy
* corneal haze or scarring
* history of corneal transplantation
* clinically active uveitis
* advanced glaucoma
* macular diseases that affect visual acuity (age-related macular degeneration, diabetic maculopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
BCVA | before and 12 months after surgery
  The change of best- corrected visual acuity
RE | 12 months after surgery
  Postoperative total refractive error
Position IOL | 1 month and 12 months after surgery
  Tilt and decentration IOL

SECONDARY OUTCOMES:
Number of complications | from day 1 until 12 months after surgery
  Rate of complications

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology Department, Military Institute of Medicine - National Research Institute, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No